CLINICAL TRIAL: NCT05270733
Title: Development of Predictive Psoriasis Response Endotypes Using Single Cell Transcriptomics in Ustekinumab Responders Versus Non-responders
Brief Title: Development of Predictive Psoriasis Response Endotypes Using Single Cell Transcriptomics
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: LEO Foundation (Unknown); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Dr. Kevin Cooper, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20220893
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
Keywords: ustekinumab; guselkumab; risankizumab; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab; guselkumab; risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Patients will be treated with ustekinumab (90mg at week 0 and week 4 by subcutaneous injection) for 8 weeks followed by treatment with guselkumab (100mg at week 0 and week 4 by subcutaneous injection) or risankizumab (150mg at week 0 and week 4 by subcutaneous injection)
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Subjects will receive ustekinumab for 8 weeks followed by guselkumab or risankizumab for 8 weeks.
  Other Names: Guselkumab; Risankizumab

SUMMARY:
The investigators propose to improve the possibility of reaching skin resolution by identifying certain markers or gene patterns that may predict patient response to certain psoriasis drugs ahead of time, thus eliminating or reducing the trial-and-error approach often employed. The ability to rule out (or in) specific therapeutics based on predictive efficacy would lead to a more personalized approach for psoriasis treatment.

To do this, the investigators will be asking participants to try two different already on the market FDA-approved psoriasis drugs for 8 weeks at a time. The investigators will be monitoring participants skin for improvements as well as taking blood and skin samples at least three times. Investigators may also ask to take stool samples and/or skin swabs.

DETAILED DESCRIPTION:
Psoriasis is a chronic systemic skin disease in which pro-inflammatory molecules contribute to the development of scaled inflamed skin and other disease-associated comorbidities such as increased risk of depression, heart attack, stroke, and metabolic syndrome. Some lesion-derived cytokines/chemokines are released into systemic circulation and increase lesional severity. Given their importance in the pathogenesis of psoriasis, the interleukins 12 (IL-12) and 23 (IL-23) are significant targets of biologic therapies.

Importantly, psoriasis patients exhibit variable responses to treatments targeting interleukins; one size does not fit all for these therapeutics. Our preliminary data demonstrates individual skin improvement (Responders) as well as lack of skin improvement (Non-Responders) in patients treated with monoclonal antibody therapy specifically targeting the shared (p40) subunit common to IL-12 and IL-23 (ustekinumab/Stelara). Interestingly, some Non-Responders to ustekinumab respond well to inhibition of the IL-23 pathway via the unique p19 subunit. We hypothesize that the pattern of differentially expressed genes (DEGs) among Responders and Non-Responders following anti-IL-12 and anti-IL-23 therapy may enable us to predict the likelihood of patient response to p40 antagonism as well as antagonism of the p19 subunit of IL-23. Single cell transcriptome analysis will be used to generate gene expression patterns that identify variable patient response patterns (endotypes).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with plaque-type psoriasis defined by either:

  * A board-certified dermatologist, OR
  * Dermatology Nurse Practitioner, OR
  * Skin punch biopsy
* Insurance that includes an anti-p40 biologic (ustekinumab/.Stelara) and at least one anti-p19 biologic (guselkumab/Tremfya or risankizumab/Skyrizi)
* Must be naive to ustekinumab, guselkumab, and risankizumab.
* Involvement of body surface area (BSA) of at least 10% at screening and baseline visit.
* Able to give informed consent under IRB approval procedures

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to get pregnant 8 weeks before, during, and 8 weeks after the study.
* Inability to provide informed consent
* Inability to secure ustekinumab and either gusekumab or risankizumab for use while on trial
* Use of tanning booths for at least 4 weeks prior to baseline visit
* Current or recent use of topical steroid, tar, phototherapy, Vitamin D, or retinoid therapy to target lesions for at least 2 weeks prior to baseline visit and for duration of trial
* Current or recent use of systemic or biologic therapy for at least 8 weeks prior to baseline visit
* Patients with psoriatic arthritis or other rheumatologic diseases (e.g., Crohn's disease).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of a unique differentially expressed gene set in patients with psoriasis that may predict disease response following antagonism to IL-12 and/or IL-23. | 24 weeks
  Single-cell RNA transcriptomics from whole blood isolate from identify unique differentially expressed gene sets in patients following antagomism to IL-12 and/or IL-23.

SECONDARY OUTCOMES:
Identification of a cell subset that is a modified and predictive of disease response following antagonism to IL-12 and/or IL-23 | 24 weeks
  Single-cell RNA sequencing or flow cytometry to identify a cell subset that is a modified and predictive of disease response following antagonism to IL-12 and/or IL-23.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cooper, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No